CLINICAL TRIAL: NCT01329185
Title: Double Blinded Placebo Controlled Study to Assess Clinical and Antiviral Activity of Valganciclovir (VAL) in Solid Organ Transplant Donors to Reduce Viral Transmission From Donor to Recipient
Brief Title: Treating Kidney Donors With Valganciclovir to Reduce Viral Transmission to Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1012M93572
Record Dates: First submitted 2011-04-01; First posted 2011-04-05 (Estimated); Results first posted 2014-06-20 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: EBV Viremia; CMV Viremia
Keywords: EBV Viremia in posttransplant kidney recipients; CMV viremia in posttransplant kidney recipients
MeSH Terms: interventions — Valganciclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Eligible consenting kidney transplant donors who are randomized to receive placebo will be given 1 placebo in morning and 1 in evening for 14 days prior to transplant date
  Interventions: Drug: Placebo
- Valganciclovir (Experimental): Eligible consenting kidney transplant donors who are randomized to the experimental arm of the study will receive 450mg of Valganciclovir twice a day for 14 days prior to the transplant date
  Interventions: Drug: Valganciclovir

INTERVENTIONS:
Drug: Valganciclovir — Valganciclovir 450mg twice a day for 14 days prior to transplant date
  Arms: Valganciclovir
Drug: Placebo — 1 capsule twice a day for 14 days prior to transplant date
  Arms: Placebo

SUMMARY:
The aim of our study is to reduce viral (CMV and EBV) transmission from donor to recipient. The discovery that anti-retroviral therapy to mothers with HIV reduced transmission of the virus to their babies was pivotal to the prevention of AIDS and so along the same lines the investigators will test the hypothesis that 14 days of the anti-viral Valganciclovir (VAL) to kidney donors prior to the transplant compared to placebo will reduce EBV and CMV viremia in the 1st year posttransplant in pediatric kidney recipients.

DETAILED DESCRIPTION:
The potency of new immunosuppressive agents has reduced the risk of the body's immune system rejecting a transplanted kidney. However, this has come with a price. Kidney transplant recipients now face a higher risk of serious infections and related malignancies.

Viral infections are a significant cause of posttransplant morbidity and mortality and two of the herpes viruses have the greatest impact: Epstein-Barr virus (EBV) and Cytomegalovirus (CMV). CMV disease can manifest posttransplant as fever, leukopenia, or mild to severe organ involvement (including pneumonitis, hepatitis, pancreatitis, colitis, meningoencephalitis, and rarely myocarditis). EBV can present posttransplant as infectious mononucleosis syndrome, hepatitis and, in the worse case scenario, a potentially fatal lymphoproliferative disorder called Post-Transplant Lymphoproliferative Disease (PTLD). Moreover, subclinical CMV and/or EBV viremia have been associated with deterioration in kidney function in kidney transplant recipients. Thus, the potential negative impact of these viruses on the lives of transplant recipients is profound and, unfortunately, the complications of these post-transplant viral infections are common and occur despite standard antiviral prophylaxis in the first year posttransplant.

These viral infections, in most instances, originate from the donor organ where these viruses reside in a dormant state, counterbalanced by the donor's healthy immune system. Upon transplantation into the recipient, whose immune system is then severely suppressed by anti-rejection drugs, these viruses become activated, often leading to the above described complications.

The aim of our study is to reduce viral (CMV and EBV) transmission from donor to recipient. The discovery that anti-retroviral therapy to mothers with HIV reduced transmission of the virus to their babies was pivotal to the prevention of AIDS and so along the same lines the investigators will test the hypothesis that 14 days of the anti-viral Valganciclovir (VAL) to kidney donors prior to the transplant compared to placebo will reduce EBV and CMV viremia in the 1st year posttransplant in pediatric kidney recipients. We aim to enroll 20 donor-recipient pairs.

ELIGIBILITY:
Inclusion criteria:

* Any person approved as a kidney transplant donor with a recipient who has never undergone a previous transplantation
* Kidney transplant donor must be 18 years old or older
* The kidney transplant donor must be positive for CMV IgG and / or EBV IgG
* The donor must be to a recipient that is discordantly seronegative for the virus for which the donor is seropositive (D+ R-)
* They must have provided signed informed consent
* The potential donors must be willing to contribute samples of blood and oral washings at regular intervals
* The potential donor must state willingness to use effective contraception during treatment and 30 days following receiving the study drug/placebo
* All females must have a negative pregnancy test
* Person must have estimated creatinine clearance (Cockcroft and Gault method) >= 60 ml/min
* Person must have Absolute neutrophil count >= 1000 cells/uL
* Person must have Platelets >= 100,000/uL
* Person must have Hemoglobin >= 9.5 g/dL

Exclusion criteria:

* Any potential kidney transplant donor who is seronegative for both CMV & EBV IgG
* Any potential kidney transplant donor who is receiving or have received anti-herpes medication in the past week
* Any potential kidney transplant donor to a recipient who has received a previous solid organ transplant
* Any potential kidney transplant donor who is immunosuppressed due to medical disease and/or immunosuppressive or immunomodulating medications
* Any potential kidney transplant donor who is breast feeding during the study
* Any potential kidney transplant donor who is on corticosteroids

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priya Verghese, MD, MPH, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Vernooij RW, Michael M, Ladhani M, Webster AC, Strippoli GF, Craig JC, Hodson EM. Antiviral medications for preventing cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2024 May 3;5(5):CD003774. doi: 10.1002/14651858.CD003774.pub5. PMID 38700045
- [Derived] Verghese PS, Evans MD, Hanson A, Hathi J, Chinnakotla S, Matas A, Balfour HH Jr. Valacyclovir or valganciclovir for cytomegalovirus prophylaxis: A randomized controlled trial in adult and pediatric kidney transplant recipients. J Clin Virol. 2024 Jun;172:105678. doi: 10.1016/j.jcv.2024.105678. Epub 2024 Apr 22. PMID 38688164

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Valganciclovir
Started | 10 | 7
CMV Disease | 1 | 0
PTLD | 1 | 0
Completed | 10 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible kidney transplant donors were enrolled at the University of Minnesota Medical Center.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Valganciclovir | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Continuous [Mean (Full Range); unit: years] — Donor Age at Transplant
  years | 43.4 [30.7 to 54.5] | 47 [29.7 to 66.6] | 44.8 [29.7 to 66.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 3 | 1 | 4
Region of Enrollment [Number; unit: participants] — Donors were recruited from the University of Minnesota Medical Center
  participants
    United States | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Incidence of EBV or CMV Related Disease in Transplant Recipient
Description: Incidence of EBV or CMV related disease in the transplant recipients of enrolled donors.
Time Frame: At least 1 year
Measure: Number; unit: participants
Arm/Group | Placebo | Valganciclovir
Number analyzed (Participants) | 10 | 7
participants | 2 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Valganciclovir
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 2/10 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Valganciclovir (N=7)
Headache (General disorders) | 1 (1) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was unblinded 2 months following the enrollment of the final donor, when a recipient developed post-transplant lymphoproliferative disorder with evidence of EBV infection at the single cell level by detection of EBV encoded small nuclear RNA.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes